CLINICAL TRIAL: NCT04931719
Title: Comparing Efficacy of Platelet-rich Plasma (PRP) Combined With Different Hyaluronan for the Treatment of Knee Osteoarthritis: a Randomized Control Trial
Brief Title: Comparing Efficacy of PRP Combined With Different Hyaluronan for the Treatment of Knee Osteoarthritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Shu-Fen Sun, MD, Neurorehabilitation Director, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VGHKS109-128
Record Dates: First submitted 2021-06-10; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Knee Osteoarthritis
Keywords: Hyaluronic acid; Knee; Osteoarthritis; Platelet-rich plasma
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: The purpose of this study was to compare the efficacy of a single Artz injection followed by PRP with a single HYAJOINT Plus injection followed by PRP in the management of knee OA.
Who Masked: Participant, Outcomes Assessor
Masking Description: One of the investigator, blinded to the allocation groups, performed all the assessments. The patients were blinded, by preventing visual access to the injection field with a screen placed between them and their knee during the injection process. They were not informed of which HA they had received during the study period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the PRP+Artz group (Active Comparator): The patients in the PRP+Artz group received one intraarticular Artz injection (2.5 ml) followed consecutively by one intraarticular injection of PRP (3ml).
  Interventions: Combination Product: PRP+Artz group; Combination Product: PRP+ HYAJOINT Plus group
- the PRP+HYAJOINT Plus group (Experimental): The patients in the PRP+HYAJOINT Plus group received one intraarticular HYAJOINT Plus injection (3ml) followed by one intraarticular injection of PRP (3ml).
  Interventions: Combination Product: PRP+Artz group; Combination Product: PRP+ HYAJOINT Plus group

INTERVENTIONS:
Combination Product: PRP+Artz group — The patients in the PRP+Artz group received one intraarticular Artz injection (2.5 ml) followed consecutively by one intraarticular injection of PRP (3ml).
Combination Product: PRP+ HYAJOINT Plus group — The patients in the PRP+HYAJOINT Plus group received one intraarticular HYAJOINT Plus injection (3ml) followed by one intraarticular injection of PRP (3ml).

SUMMARY:
Either PRP or HA is each effective for treating knee OA. However, the efficacy of combined PRP and HA injections remains unknown clinically.

DETAILED DESCRIPTION:
Intraarticular plasma-rich platelet (PRP) or hyaluronic acid (HA) was each effective for knee osteoarthritis(OA). The efficacy of combined injections remains unknown. This study aimed to evaluate the efficacy of PRP combined with different hyaluronan for treating knee OA. In a prospective, randomized-controlled trial, 95 patients with Kellgren-Lawrence grade 2 knee OA were randomized to receive a single intraarticular Artz (10mg/ml) followed by PRP (N=48) into target knee or single HYAJOINT Plus (20mg/ml) injection followed by PRP (N=47). Primary outcome was the change from baseline in the visual analog scale (VAS) pain at 6 months. Secondary outcomes included the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Lequesne index, single leg stance test (SLS), use of rescue analgesics and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age of 20-85 years Symptomatic knee osteoarthritis for more than 6 months despite analgesics, NSAIDs, or physical therapy Kellgren-Lawrence grade-2 knee osteoarthritis seen on radiographs made within previous 6 months Radiological evidence of bilateral knee OA was accepted if global pain VAS in the contralateral knee was less than 30 mm.

Exclusion Criteria:

* Previous orthopedic surgery on spine or lower limb Disabling osteoarthritis of either hip or foot Knee instability, apparent joint effusion, or marked valgus/varus deformity Known allergy to avian proteins or hyaluronan products Confirmed or suspected pregnancy, or lactating Intra-articular injections into knee in previous 6 months Any specific medical conditions (rheumatoid arthritis, active infection, hemiparesis, neoplasm, hematological etc.) that would interfere with assessments

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
visual analog scale (VAS) pain change | Month 6
  the change from baseline in the visual analog scale (VAS) pain score at 6 months. The patient rated the average severity of knee pain on knee movement over the previous week on a 0-100 mm VAS (0 = no pain to 100 = worst possible pain)

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC, Likert Scale), t | Month 6
  (WOMAC, Likert Scale) is a 24-item questionnaire with 3 subscales measuring pain, stiffness, and physical function. Total score is 96 and higher scores indicate worse outcomes.
the Lequesne index | Month 6
  Lequesne index was used to assess severity of knee symptoms during the last week. It includes the measurement of pain, walking distance, and activities of daily living. Maximal score is 24 and higher scores represent worse function.
single-leg stance test (SLS) | Month 6
  Single-leg stance test (SLS) is done by raising one foot up without touching it to the supported lower extremity with target knee and maintain balance for as long as possible. Each participant performed 3 trials, and the best result of the 3 trials was recorded.
patient satisfaction. | Month 6
  Patients were asked to rate their treatment satisfaction compared to the preinjection condition, using a 100 mm VAS (0= completely dissatisfied, 100=completely satisfied).
consumption of analgesics | Month 6
  Acetaminophen (500mg; maximum daily dose, 4 g) was the only rescue medication allowed for knee pain during the study period, Use of rescue medication during the study period was recorded in a patient diary.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Fen Sun, Principal Investigator — Department of Physical Medicine and Rehabilitation, Kaohsiung Veterans General Hospital
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sun SF, Lin GC, Hsu CW, Lin HS, Liou IS, Wu SY. Comparing efficacy of intraarticular single crosslinked Hyaluronan (HYAJOINT Plus) and platelet-rich plasma (PRP) versus PRP alone for treating knee osteoarthritis. Sci Rep. 2021 Jan 8;11(1):140. doi: 10.1038/s41598-020-80333-x. PMID 33420185
- [Result] Sanchez M, Anitua E, Delgado D, Sanchez P, Prado R, Orive G, Padilla S. Platelet-rich plasma, a source of autologous growth factors and biomimetic scaffold for peripheral nerve regeneration. Expert Opin Biol Ther. 2017 Feb;17(2):197-212. doi: 10.1080/14712598.2017.1259409. Epub 2016 Nov 28. PMID 27845852
- [Result] Laudy AB, Bakker EW, Rekers M, Moen MH. Efficacy of platelet-rich plasma injections in osteoarthritis of the knee: a systematic review and meta-analysis. Br J Sports Med. 2015 May;49(10):657-72. doi: 10.1136/bjsports-2014-094036. Epub 2014 Nov 21. PMID 25416198
- [Result] Jain NK, Gulati M. Platelet-rich plasma: a healing virtuoso. Blood Res. 2016 Mar;51(1):3-5. doi: 10.5045/br.2016.51.1.3. Epub 2016 Mar 25. No abstract available. PMID 27104183
- [Result] Mlynarek RA, Kuhn AW, Bedi A. Platelet-Rich Plasma (PRP) in Orthopedic Sports Medicine. Am J Orthop (Belle Mead NJ). 2016 Jul-Aug;45(5):290-326. PMID 27552452
- [Result] Webb D, Naidoo P. Viscosupplementation for knee osteoarthritis: a focus on Hylan G-F 20. Orthop Res Rev. 2018 Oct 23;10:73-81. doi: 10.2147/ORR.S174649. eCollection 2018. PMID 30774462
- [Result] Sun SF, Hsu CW, Lin HS, Liou IH, Chen YH, Hung CL. Comparison of Single Intra-Articular Injection of Novel Hyaluronan (HYA-JOINT Plus) with Synvisc-One for Knee Osteoarthritis: A Randomized, Controlled, Double-Blind Trial of Efficacy and Safety. J Bone Joint Surg Am. 2017 Mar 15;99(6):462-471. doi: 10.2106/JBJS.16.00469. PMID 28291178
- [Result] Russo F, D'Este M, Vadala G, Cattani C, Papalia R, Alini M, Denaro V. Platelet Rich Plasma and Hyaluronic Acid Blend for the Treatment of Osteoarthritis: Rheological and Biological Evaluation. PLoS One. 2016 Jun 16;11(6):e0157048. doi: 10.1371/journal.pone.0157048. eCollection 2016. PMID 27310019
- [Result] Weibrich G, Hansen T, Kleis W, Buch R, Hitzler WE. Effect of platelet concentration in platelet-rich plasma on peri-implant bone regeneration. Bone. 2004 Apr;34(4):665-71. doi: 10.1016/j.bone.2003.12.010. PMID 15050897
- [Result] McConnell S, Kolopack P, Davis AM. The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC): a review of its utility and measurement properties. Arthritis Rheum. 2001 Oct;45(5):453-61. doi: 10.1002/1529-0131(200110)45:53.0.co;2-w. No abstract available. PMID 11642645
- [Result] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Result] Lequesne MG, Mery C, Samson M, Gerard P. Indexes of severity for osteoarthritis of the hip and knee. Validation--value in comparison with other assessment tests. Scand J Rheumatol Suppl. 1987;65:85-9. doi: 10.3109/03009748709102182. PMID 3479839
- [Result] Srinivasan PP, McCoy SY, Jha AK, Yang W, Jia X, Farach-Carson MC, Kirn-Safran CB. Injectable perlecan domain 1-hyaluronan microgels potentiate the cartilage repair effect of BMP2 in a murine model of early osteoarthritis. Biomed Mater. 2012 Apr;7(2):024109. doi: 10.1088/1748-6041/7/2/024109. Epub 2012 Mar 29. PMID 22455987
- [Result] Abate M, Verna S, Schiavone C, Di Gregorio P, Salini V. Efficacy and safety profile of a compound composed of platelet-rich plasma and hyaluronic acid in the treatment for knee osteoarthritis (preliminary results). Eur J Orthop Surg Traumatol. 2015 Dec;25(8):1321-6. doi: 10.1007/s00590-015-1693-3. Epub 2015 Sep 24. PMID 26403468
- [Result] Zhao J, Huang H, Liang G, Zeng LF, Yang W, Liu J. Effects and safety of the combination of platelet-rich plasma (PRP) and hyaluronic acid (HA) in the treatment of knee osteoarthritis: a systematic review and meta-analysis. BMC Musculoskelet Disord. 2020 Apr 11;21(1):224. doi: 10.1186/s12891-020-03262-w. PMID 32278352
- [Derived] Huang HY, Hsu CW, Lin GC, Lin HS, Chou YJ, Liou IH, Sun SF. Comparing efficacy of a single intraarticular injection of platelet-rich plasma (PRP) combined with different hyaluronans for knee osteoarthritis: a randomized-controlled clinical trial. BMC Musculoskelet Disord. 2022 Nov 4;23(1):954. doi: 10.1186/s12891-022-05906-5. PMID 36329428